CLINICAL TRIAL: NCT04244097
Title: The Evaluation of the Analgesic Effect of Intraperitoneal Bupivacaine Versus Bupivacaine With Neostigmine on Postoperative Pain in Laparoscopic Cholecystectomy:A Prospective, Randomized, Comparative, Double-blind Study.
Brief Title: The Effect of Intraperitoneal Bupivacaine Versus Bupivacaine With Neostigmine on Pain in Laparoscopic Cholecystectomy
Acronym: RCTcompstud
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Sara Farouk Kassem Habib, lecturer of anesthesiology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-273-2019
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Neostigmine

STUDY DESIGN:
Intervention Model Description: * Group 1 (Bupivacaine group= B group) will receive a 50 mL solution of bupivacaine 0.25% intraperitoneal instilled solution.
  * Group 2 (Bupivacaine neostigmine group=BN group) will receive 500 μg neostigmine mixed with bupivacaine 0.25% with a total volume of 50 mL intraperitoneal instilled solution.
Who Masked: Care Provider
Masking Description: Patients will be randomly allocated to one of two groups with the help of computer generated random number tables in opaque sealed envelopes prepared by an anaesthesiologist not part of the study. The envelops will be opened by the staff nurse, and peritoneal solution will be prepared according to group allocation by anaesthesiologist who is not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- B group (Experimental): -Group 1 (Bupivacaine group= B group) will receive a 50 mL solution of bupivacaine 0.25% intraperitoneal instilled solution.
  Interventions: Drug: Bupivacaine Hydrochloride
- BN group (Active Comparator): Group 2 (Bupivacaine neostigmine group=BN group) will receive 500 μg neostigmine mixed with bupivacaine 0.25% with a total volume of 50 mL intraperitoneal instilled solution.
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Neostigmine

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — after induction of general anesthesia and before the start of surgery, after inflating the pneumoperitoneum and before any surgical manipulation, the surgeon infuse 50 mL of blinded solution (bupivacaine or bupivacaine neostigmine) intraperitoneally to the sub-diaphragmatic space and gall bladder area guided by the camera and the patients are kept in Trendelenburg position for 5-10 minutes. Thereafter all patients will be positioned in the anti-Trendelenburg position to start the surgery and the laparoscopic procedure will be carried out in a standard fashion.
  Other Names: Marcaine
Drug: Neostigmine — after induction of general anesthesia and before the start of surgery, after inflating the pneumoperitoneum and before any surgical manipulation, the surgeon infuse 50 mL of blinded solution (bupivacaine or bupivacaine neostigmine) intraperitoneally to the sub-diaphragmatic space and gall bladder area guided by the camera and the patients are kept in Trendelenburg position for 5-10 minutes. Thereafter all patients will be positioned in the anti-Trendelenburg position to start the surgery and the laparoscopic procedure will be carried out in a standard fashion.
  Other Names: prostigmin
  Arms: BN group

SUMMARY:
Injection of intraperitoneal bupivacaine revealed an analgesic effect whether injected alone or in combination with other adjuvants, which increase duration of analgesia and decrease the dose of administered bupivacaine thus minimizing its side effects e.g. Opioids, Corticosteroids and Magnesium sulphate.

Neostigmine, a cholinesterase inhibitor that produces muscarinic receptor-mediated analgesia, increased postoperative analgesia when combined with local anaesthetics. Peripheral afferent nerve fibres contain muscarinic receptors, these could be a good target for pain suppression.

DETAILED DESCRIPTION:
The use of neostigmine as adjuvant to intraperitoneal bupivacaine was not previously investigated. In this study the investigators will compare the analgesic effect of bupivacaine alone and bupivacaine in combination with neostigmine when injected intraperitoneal in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* • American Society of Anaesthesiologist (ASA) I-II.

  * Age 18 - 60 years.
  * Elective laparoscopic cholecystectomy.
  * Body Mass Index (BMI) <35 (kg/m2).

Exclusion Criteria:

* • Anaphylaxis to local anaesthetics.

  * Anaphylaxis to Neostigmine.
  * American Society of Anaesthesiologist (ASA) III-IV.
  * Chronic pain diseases.
  * Acute cholecystitis.
  * Psychological or nervous system diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Time of first analgesic requirements (in hours) after extubation | 24 Hours post-operatively.
  hours

SECONDARY OUTCOMES:
• Total dose of intravenous pethidine (mg/24 hours). | 24 hours
  milligram
• The use of intra-operative rescue analgesia. | intraoperative period
  milligram
• The severity of post-operative shoulder pain assessed by visual analogue scale | 24 Hours post-operatively.
  segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain 0 (no pain), 10(worst pain). The common format is a horizontal bar or line
• The severity of post-operative abdominal pain assessed by visual analogue scale | 24 hours posoperatively
  segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain 0 (no pain), 10(worst pain). The common format is a horizontal bar or line
• Post-operative nausea and vomiting assessed by postoperative nausea and vomiting score | 24 hours postoperatively
  A simplified risk score for predicting postoperative nausea and vomiting female gender, history of PONV and/or motion sickness, non-smoking status, and postoperative use of opioids. When 0, 1, 2, 3, or 4 factors are present, the risk of postoperative nausea and vomiting is 10%, 20%, 40%, 60%, or 80%, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Sara Fa Habib, PhD, Principal Investigator — Kasr El Aini -Faculty Of Medicine- Cairo University
Locations (1):
- Sara Farouk Kassem Habib, Cairo, El Azbakeya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
results of the study or medical data like vital signs only could be shared
Supporting Information: Study Protocol, SAP
Time Frame: 2 months after publication
Access Criteria: data concerning results charts will be available by contacting principal investigator

REFERENCES:
- [Result] Khurana S, Garg K, Grewal A, Kaul TK, Bose A. A comparative study on postoperative pain relief in laparoscopic cholecystectomy: Intraperitoneal bupivacaine versus combination of bupivacaine and buprenorphine. Anesth Essays Res. 2016 Jan-Apr;10(1):23-8. doi: 10.4103/0259-1162.164731. PMID 26957685
- [Result] LAURETTI G. Postoperative analgesia by intra-articular and epidural neostigmine following knee surgery. Reg Anesth Pain Med [Internet]. 1999 Jun;24(3):17.